CLINICAL TRIAL: NCT01296048
Title: Verify the Functions and Efficiency of Transtek Glass Body Analyzer, GBF-830, GBF-835, GBF-950, SA-15
Brief Title: Clinical Test for Transtek Glass Body Analyzer
Acronym: GBA
Status: Completed | Type: Observational
Sponsor: Leo Wang (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Leo Wang, Team Leader, BTS International
Organization: BTS International (Other)
Other Study IDs: Transtek GBA; BTS-TRANS02 (Other: BTSInternational)
Record Dates: First submitted 2011-02-12; First posted 2011-02-15 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Weight; Body Fat Disorder; Bone Mass
Keywords: weight; body fat; total body water; bone mass; muscle mass
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Body Analysis
  Interventions: Device: Comparison test

INTERVENTIONS:
Device: Comparison test — Scaleman Body Fat Scales, FS-148BW1, accuracy: ±0.1kg and range: 0-180kg.
  Other Names: Brand names: Scaleman; Serial numbers: SBFS1002-351; Code name: FS-148BW1

SUMMARY:
The clinical protocol of the clinical testing of this device:

1. Objective of the test: To verify the functions and efficiency of devices.
2. Test methods and procedures: Comparison Test.
3. DUT: Transtek Glass Body Analyzer, Model: GBF-830, GBF-835, GBF-950, and SA-15.
4. Comparison device: Scaleman Body Fat Scales, FS-148BW1 (Predicate Device).
5. Study endpoints: Transtek devices and the predicate device are substantial equivalence.
6. Statistical methodology used: Description of statistical methods.
7. Result: Efficiencies of Transtek devices and predicate device are in the same level.

DETAILED DESCRIPTION:
Hospital Information The data was collected by West China Medical College Clinical Investigator Team at Wuhou District Hospital, No. 9 Tongzilin Road, Wuhou District, Chengdu 610041, P. R. China.

Investigator: Catharine Zhang, Nurse A; Vivian Luo, Nurse B; Dr. James Zhu, Sponsor.

Contact Dr. James Zhu Tel: +86 1330 8036568 Used Equipments DUT (Device Under Test): Transtek Glass Body Analyzer, GBF-830, GBF-835, GBF-950, and SA-15.

Reference Device: Scaleman Body Fat Scales, FS-148BW1 (Predicate Device). Test Protocol

1. Test Purpose:

   The aim of clinical test is to collect weight, body fat, total body water, bone mass, and muscle mass reading value which measured by DUT and reference device.

   Note: GBF-835 has not total body water, bone mass, and muscle mass functions. So it just collects weight and body fat data.
2. Target Subject:

   The subject database shall contain at least 25 male and 25 female subjects and all above 18 years old. Patient's population analysis is bellow.
3. Test procedures 1) Record the name, age, gender, and height of each subject. 2) Let subject seated calmly for two minutes before test, dry the feet. 3) Use device to measure weight, body fat, total body water, bone mass, and muscle mass; record reading value.

4) For each subject, repeat 3) to get 3 pairs measurements. 5) Repeat step 1) to 4) for every device (DUT: GBF-830, GBF-835, GBF-950, and SA-15; and reference device: FS-148BW1).

6) Repeat step 1) to 5) for each subject. 5. Note:

1. No motion and speaking are allowed during the measurement.
2. All DUT use the same algorithms, have the same number of electrodes and contact the patient at the same body locations (feet), and operate on the same frequency.
3. Test environment: Temperature: 20±1℃; Relative humidity: 40~50%.

ELIGIBILITY:
Inclusion Criteria:

* male,female

Exclusion Criteria:

* below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population included patients whose age is above 18 years old. Male or Female.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Verify the accuracy of measure functions of device | 10 days
  Verify the functions and efficiency of these devices compare with a specified product.

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Li, Director, Principal Investigator — Wuhou District Hospital
Locations (1):
- Wuhou District Hospital, Chengdu, Sichuan, China